CLINICAL TRIAL: NCT03727100
Title: A Prospective, Multicenter, Randomized, Double-Blinded, Sham-Control Study to Evaluate the Efficacy and Safety of Clonidine Micropellets for the Treatment of Pain Associated With Lumbosacral Radiculopathy in Adults
Brief Title: Treatment of Pain Associated With Lumbosacral Radiculopathy in Adults
Acronym: RePRIEVE-CM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sollis Therapeutics, Inc. (Industry)
Collaborators: Lotus Clinical Research, LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STX-015-18-01
Record Dates: First submitted 2018-10-30; First posted 2018-11-01 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Lumbosacral Radiculopathy
MeSH Terms: interventions — salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: Clonidine Micropellet vs Sham-Control
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double-Blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Clonidine Micropellets (Active Comparator): single dose injection into the lumbar epidural space
  Interventions: Combination Product: Clonidine Micropellets
- Sham Control (Sham Comparator): non-epidural needle placement
  Interventions: Other: Sham

INTERVENTIONS:
Combination Product: Clonidine Micropellets — Injection
  Arms: Clonidine Micropellets
Other: Sham — Injection
  Arms: Sham Control

SUMMARY:
This study will evaluate the safety and effectiveness of a new pain medication in development, clonidine micropellet. Participants will receive a single injection of either clonidine micropellet or sham injection for the treatment of low back and leg pain from sciatica.

ELIGIBILITY:
Main Inclusion Criteria:

1. Be between 18 and 70 years of age (inclusive) at time the Informed Consent Form (ICF) is signed.
2. Diagnosis of unilateral radicular leg pain.
3. Women of childbearing potential must have a negative pregnancy test at Screening and within 24 hours prior to procedure and commit to adequate birth control during the the study.
4. Understands the purpose and any risks associated with the procedure required for the study and is willing to participate in the study.
5. Agrees to follow study-specific medication requirements.
6. Be able to read, write, understand, and complete study-related tasks, and adequately communicate in English.
7. Subject must have failed at least one conservative therapy in two different categories.

Main Exclusion Criteria:

1. Medical condition or radiographic evidence that, in the Investigator's opinion, could adversely impact study outcomes.
2. Received an lumbar epidural steroid injection, nerve block or similar procedure during the 4 weeks prior to Screening.
3. Female subjects who are pregnant or breastfeeding.
4. History of lumbar surgery.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2020-03-05 (Actual); Study Completion 2020-07-18 (Actual)

PRIMARY OUTCOMES:
Pain Intensity Difference (PID) for the average pain Numeric Rating Scale (NRS) from baseline to D30 in radicular leg pain | Baseline to day 60
  Difference in average pain score, using a scale of 0-10 with 0 no pain and 10 worst possible pain, from baseline to day 30.

SECONDARY OUTCOMES:
Change in Oswestry Disability Index (ODI) score | Baseline to day 30
  6 categories of 10 question, each question is scored from 0-5 (minimum to maximum). The scores range from 0-100% with lower scores meaning less disability.
Change in Numeric Rating Scale (NRS) leg pain 24 hrs post injection. | 1 day post injection
  Difference in average pain score, using a scale of 0-10 with 0 no pain and 10 worst possible pain, from injection to 24 hrs post injection.
Difference in Rescue medication consumption | Baseline to day 30
  Consumption from baseline through day 30
Percent of subjects with significant improvement in pain | Baseline to day 30
  50 percent improvement in pain from baseline to day 30

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Gilligan, MD, Principal Investigator — Brigham and Women's Hospital
Locations (33):
- United States (33):
  - Sollis Clinical Study Site 36, Mobile, Alabama
  - Sollis Clinical Study Site #41, Phoenix, Arizona
  - Sollis Clinical Study Site #44, Phoenix, Arizona
  - Sollis Clinical Study Site 29, Scottsdale, Arizona
  - Sollis Clinical Study Site 40, Tucson, Arizona
  - Sollis Clinical Study Site 49, Rancho Mirage, California
  - Sollis Clinical Study Site 28, Santa Rosa, California
  - Sollis Clinical Study Site 30, Washington D.C., District of Columbia
  - Sollis Clinical Study Site 35, Fort Lauderdale, Florida
  - Sollis Clinical Study Site 38, Miami, Florida
  - Sollis Clinical Study Site 12, Bloomington, Illinois
  - Sollis Clinical Study Site 13, Chicago, Illinois
  - Sollis Clinical Study Site 14, Kansas City, Kansas
  - Sollis Clinical Study Site, Overland Park, Kansas
  - Sollis Clinical Study Site 10, Edgewood, Kentucky
  - Sollis Clinical Study Site 16, Boston, Massachusetts
  - Sollis Clinical Study Site 15, Brookline, Massachusetts
  - Sollis Clinical Study Site 17, Shrewsbury, New Jersey
  - Sollis Clinical Study Site 25, Albany, New York
  - Sollis Clinical Study Site 31, Rochester, New York
  - Sollis Clinical Study Site 18, Winston-Salem, North Carolina
  - Sollis Clinical Study Site 21, Cleveland, Ohio
  - Sollis Clinical Study Site 33, Cleveland, Ohio
  - Sollis Clinical Study Site 19, Edmond, Oklahoma
  - Sollis Clinical Study Site 46, Eugene, Oregon
  - Sollis Clinical Study Site, Dallas, Texas
  - Sollis Clinical Study Site 34, Houston, Texas
  - Sollis Clinical Study Site 22, San Antonio, Texas
  - Sollis Clinical Study Site 43, The Woodlands, Texas
  - Sollis Clinical Study Site 20, Tyler, Texas
  - Sollis Clinical Study Site 47, Salt Lake City, Utah
  - Sollis Clinical Study Site 23, Morgantown, West Virginia
  - Sollis Clinical Study Site 27, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No